CLINICAL TRIAL: NCT01672736
Title: A Phase 1/2 Trial of ASP7487 OSI-906)in Combination With Bortezomib and Dexamethasone for the Treatment of Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: A Trial of ASP7487 (OSI-906) in Combination With Bortezomib for the Treatment of Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to stop further manufacture the study drug 'Linsitinib' in Nov 2015.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Multiple Myeloma Research Consortium (Network); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMHOSI906-MM001
Record Dates: First submitted 2012-08-01; First posted 2012-08-27 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or relapse/refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ASP7487, Velcade, Dexamethasone (Experimental): ASP7487 administered orally 75, 100 and 150 mg) BID continuously for each cycle. Bortezomib administered at 1.3 mg/m2 twice weekly for the first 8 21 day cycles and once weekly beyond cycle 9 for 35 day cycles. Dexamethasone is administered on bortezomib administration days at 20 mg
  Interventions: Drug: ASP7487, Velcade, Dexamethasone

INTERVENTIONS:
Drug: ASP7487, Velcade, Dexamethasone — ASP7487- Oral (75, 100, 150 mg)BID Bortezomib- 1.3 mg/m2 IV on days 1, 4, 8, 15 of each 21 day cycle up to cycle 8 and days 1, 5, 15, 22 of each 35 day cycle beyond cycle 9 Dexamethasone- 20 mg on the day of Bortezomib administration
  Other Names: ASP7487; Bortezomib; Dexamethasone

SUMMARY:
This is a multi-center, open-label, non-randomized study. Patients will receive ASP7487 (OSI-906) in combination with bortezomib and dexamethasone. Phase 1 involves dose escalation of the combination, whereas Phase 2 involves the expansion of ASP7487 (OSI-906) combined with bortezomib and dexamethasone at the MTD to establish the ORR. This trial will accrue patients with relapsed or relapsed/refractory MM - a disease state for which bortezomib is approved to treat by the FDA and Health Canada. The combination of ASP7487 (OSI-906) with bortezomib is supported by pre-clinical work in MM in which the combination with an IGF1-R inhibitor enhances anti-tumor activity of bortezomib.

DETAILED DESCRIPTION:
The Phase 1 portion of the study will determine the MTD and DLTs of bortezomib administered on days 1, 4, 8 and 11 of a 21-day cycle combined with ASP7487 (OSI-906) dosed twice daily orally continuously. The combination of ASP7487 (OSI-906) with bortezomib has not previously been tested. The active agent bortezomib will be used during Cycle 1 - 8 at the recommended treatment dose of 1.3 mg/m2 days 1, 4, 8 and 11 and Cycles 9+ on days 1, 8, 15 and 22 of a 5-week cycle and ASP7487 (OSI-906) will be dose escalated form 75 mg to 150mg utilizing 3+3 design

ELIGIBILITY:
Inclusion Criteria

1. Males or females, age 18 years or older.
2. Relapsed or relapse/refractory MM with at least 1 prior line of therapy for phase 1 and 1 to 5 prior lines of therapy for phase 2.
3. Patients with measurable disease defined as at least one of the following

   1. Serum M-protein ≥ 0.5 g/dl (≥ 5 g/l)
   2. Urine M-protein ≥ 200 mg/24 h
   3. Serum free light chains (FLC) assay: Involved FLC level ≥ 10 mg/dl (≥ 100 mg/l) and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
   4. Biopsy proven plasmacytoma. Prior biopsy is acceptable.
   5. If the serum protein electrophoresis is unreliable for routine M-protein measurement, quantitative immunoglobulin levels on nephrolometry or turbidometry will be followed.
4. ECOG ≤ 2 OR Karnofsky ≥ 60%.
5. Predose mean QTc≤ 450 msec or QTcF ≤ 450 msec.
6. Negative pregnancy test for Females of childbearing potential.
7. Voluntary, written informed consent.
8. Ability to understand the purpose and risks of the study.
9. Must be able to take and retain oral medications.
10. Inclusion Clinical Laboratories Criteria

    1. Absolute neutrophil count (ANC) > 1,000 cells/dL (1.0 x 109/L)
    2. Platelet count > 50,000 cells/dL (50 x 109/L)
    3. Hemoglobin ≥ 8.0 g/dL (4.96 mmol/L)
    4. Serum AST or ALT ≤ 1.2 x ULN
    5. Total bilirubin within normal limits
    6. Creatinine clearance ≥ 30 mL/min
    7. Serum creatinine ≤ 1.5 x ULN
    8. Serum calcium (ionized or corrected for albumin) ≥ 2.0 mmol/L (8.0 mg/dL or 1.0 mmol/L ionized calcium) to ≤ 1.2 x ULN.
    9. Serum potassium, and magnesium within normal limits
    10. HgbA1c of ≤ 7%
    11. Troponin I or T within normal limits
    12. BNP or NT-proBNP within normal limits
    13. Fasting glucose of ≤126 mg/dL (7.0 mmol/L).
11. Resolution of prior treatment associated toxicities to ≤ grade 1

Exclusion Criteria

1. Bortezomib refractory patients are not permitted on the Phase 2 part of the study.
2. Diagnosed or treated for another malignancy within 3 years of enrollment, except completely resected basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
3. Patient has received other investigational drugs or chemotherapy within 21 days or approved anti-myeloma therapy within 14 days.
4. History (within the last 6 months) of significant cardiovascular disease.
5. Mean QTcF interval > 450 msec at screening.
6. Prior autologous, peripheral stem cell transplant within 12 weeks of the first dose of study drug.
7. Daily requirement for corticosteroids (except for inhalation corticosteroids).
8. Patients with evidence of mucosal or internal bleeding and/or platelet transfusion refractory (i.e., unable to maintain a platelet count ≥ 50,000 cells/dL).
9. Known active infection requiring parenteral or oral anti-infective treatment.
10. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation.
11. Use of any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient.
12. Patient has hypersensitivity to any of the components of study drugs.
13. Known HIV or active hepatitis B or C viral infection.
14. Diabetes mellitus currently requiring insulin or insulinotropic therapy or prior history of steroid induced diabetes.
15. History of cerebrovascular accident (CVA) within 6 months prior to registration or that is not stable.
16. Prior therapy with an IGF-1R inhibitor.
17. Use of drugs that have a risk of causing QT interval prolongation and/or have a known risk of causing Torsades de Pointes (TdP) before 14 days or the recommended 5 half-life.
18. Use of strong/moderate CYP1A2 inhibitors.
19. Gastro-intestinal abnormalities that could affect the absorption of study drug.
20. Peripheral neuropathy ≥ grade 2.
21. Significant liver disease or metastatic disease to the liver
22. History of amyloid, plasma cell leukemia or CNS involvement.
23. Radiation therapy or major surgical procedure within 4 weeks of the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-09; Primary Completion 2017-03-27 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Trudel, MD, Principal Investigator — UHN-PMH
Locations (6):
- United States (2):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University Of Chicago Medical Center, Chicago, Illinois
- Canada (4):
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Sir Mortimer B. Davis-Jewish General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment under this IND was stopped prematurely due to the drug manufacturer's decision to terminate the development of the study drug, Linsitinib (letter dated 1 November 2015). Therefore, the study did not proceed to Phase II portion of the study protocol. The available study drug supply at the study sites expired on 31 May 2016.
Period: Overall Study
Arm/Group | ASP7487, Velcade, Dexamethasone
Started | 19 (Phase I study part stopped early due to manufacturer's decision to stop further drug development.)
Completed (Phase II part of the study not done due to termination of further study drug development.) | 16 (3 patients taken off study due to non-availability of further study (Linsitinib) drug supply.)
Not Completed | 3
Not completed — Available drug expired on 31 May 16 | 3

BASELINE CHARACTERISTICS:
Arm/Group | ASP7487, Velcade, Dexamethasone
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 18
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of the Combination of ASP7487 (OSI-906) With Velcade and Dexamethasone
Description: * Phase 1: To determine the maximum tolerated dose (MTD) of ASP7487 (OSI-906) administered in combination with the recommended dose and schedule of bortezomib and dexamethasone;
  * Phase 2: To evaluate the antitumor activity of ASP7487 (OSI-906) in combination with bortezomib and dexamethasone at the MTD established from the Phase 1 component.
Time Frame: 45 months
Measure: Number; unit: milligrams
Arm/Group | ASP7487, Velcade, Dexamethasone
Number analyzed (Participants) | 19
milligrams
  Linsitinib starting dose in milligrams | 75
  Linsitinib maximum dose in milligrams | 150

ADVERSE EVENTS:
Time Frame: 4 years and 10 months. This period includes the time period from study activation to the final data analysis, the results of which are presented here.The adverse event data was collected from study activation on 3 Oct 2012 up to 22 Aug 2017.
Description: Adverse Events were graded in accordance with CTCAE v4.03
Arm/Group | ASP7487, Velcade, Dexamethasone
All-Cause Mortality (participants affected / at risk) | 2/19
Serious Adverse Events (participants affected / at risk) | 8/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP7487, Velcade, Dexamethasone (N=19)
Alanine Aminitransferase Increased (Investigations) | 1 (1)
Asparate Aminotransferase increased (Investigations) | 1 (1) — Occured in the same patient with increased Alanine Aminotransferase
Delirium (Nervous system disorders) | 1 (1) — not related to study drug
Lung infection (Infections and infestations) | 2 (2)
Death due to multiple myeloma (General disorders) | 1 (1) — Death due to progressive disease
Cardiac arrest (Cardiac disorders) | 1 (1) — Probably related to bortezomib
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
fever (General disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASP7487, Velcade, Dexamethasone (N=19)
Anemia (Blood and lymphatic system disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 7
Pneumonia/influenza (Infections and infestations) | 4
Creatinine Increased (Investigations) | 8
Platelet count decreased (Investigations) | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Neuropathy (Nervous system disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6

LIMITATIONS AND CAVEATS:
Patient enrollment was stopped prematurely due to the drug manufacturer's decision to terminate the development of the study drug, Linsitinib. The study did not proceed to Phase II portion of the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT01672736/Prot_SAP_000.pdf